CLINICAL TRIAL: NCT05412589
Title: Intravenous mFOLFOX7 Plus Camrelizumab and Apatinib for CNLC Stage III Hepatocellular Carcinoma
Brief Title: mFOLFOX7 Plus Camrelizumab and Apatinib for Advanced HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2021-KY-139
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Stage III Hepatocellular Cancer (CNLC Staging)
MeSH Terms: conditions — Liver Neoplasms | interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intravenous mFOLFOX7 combined with Camrelizumab and apatinib (Experimental): Combination of systemic chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin (mFOLFOX7) , targeted drugs (Apatinib 250mg), and anti-PD-1 immunotherapy (Camrelizumab 200mg)
  Interventions: Drug: mFOLFOX7+Camrelizumab+Apatinib

INTERVENTIONS:
Drug: mFOLFOX7+Camrelizumab+Apatinib — Drug: Leucovorin 200mg/m2 administered IV on Days 1 of a 21 day cycle Drug: Oxaliplatin 85 mg/m2 IV on Days 1 of a 21 day cycle. Drug: Fluorouracil 5-FU continuous infusion: 400mg/m2 on D1 and then 2400mg/m2 for 46h of each 21 day cycle.
  Drug: Camrelizumab 200mg infusion on D1 for every 21 days Drug: Apatinib 250mg，po，qd for every 21 days
  Other Names: Combination Product: Systemic chemotherapy combined with Apatinib and Camrelizumab

SUMMARY:
This is a prospective, one-arm, phase II clinical study of intravenous mFOLFOX6 plus Camrelizumab combined with apatinib for CNLC stage III hepatocellular carcinoma

DETAILED DESCRIPTION:
The combination of anti-angiogenesis and immune checkpoint blockade showed promising outcomes for advanced HCC. Hepatic artery infusion chemotherapy （HAIC） combined with apatinib and camrelizumab could augment treatment efficacy in preliminary study. But HAIC had disadvantages such as technical limitations, expensive cost and poor patient comfort. In the present study, we aimed to investigate the efficacy and safety of Venous Infusion Chemotherapy（VIC） plus camrelizumab and apatinib for CNLC stage Ⅲ HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study and signed informed consent;
2. Age 18-75, male or female;
3. ECOG PS score 0-2;
4. Child-pugh liver function grading: Grade A or B
5. The clinical diagnosis conforms to primary hepatocellular carcinoma (HCC) and the lesion conforms to stage III according to China liver cancer staging (CNLC)
6. Did not received any type of other first-line drugs such as Sorafenib
7. According to RECIST 1.1 standard, patients have at least one measurable lesion (CT/MRI scan long diameter ≥10mm or CT/MRI scan short diameter ≥15mm for lymph node lesions, and the lesion has not received radiotherapy, freezing or other local treatments);
8. Expected survival ≥ 12 weeks;
9. The function of vital organs meets the following requirements (excluding the use of any blood component and cell growth factor within 14 days) :

   Blood routine:

   White blood cells count ≥3.0×109/L Platelet count ≥70×109/L Hemoglobin ≥80g/L;

   Liver and kidney function:

   Serum creatinine (SCr) ≤ 1.5 times upper limit of normal value (ULN) or creatinine clearance ≥50 ml/min (Cockcroft-Gault formula); Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); AST or ALT levels ≤ 3 times the upper limit of normal value (ULN)
10. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during and within six months of the end of medication;Patients with negative serum or urine pregnancy tests within 7 days prior to study inclusion and who must be non-lactating, and males should agree to use contraceptives during the study period and for 6 months after the end of the study period.
11. Subjects have good compliance and cooperate with the follow-up.
12. Subjects with HBV or HCV infection should receive anti-virus treatment without interfron.

Exclusion Criteria:

1. Have received immunotherapeutic drugs or interferon in the past.
2. Severe allergic reaction to other monoclonal antibodies.
3. Female subjects with pregnancy.
4. Patients with congenital or acquired immune deficiencies.
5. Abnormal coagulation function (INR>2.0, PT>16s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy, and allow preventive use of low-dose aspirin and low-molecular-weight heparin
6. The patient has suffered from other malignant tumors at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ)
7. The patient has active infection, fever of unknown origin within 7 days (CTCAE>2)
8. Patients with congenital or acquired immune deficiencies.
9. With clinical symptoms or diseases of the heart that are not well controlled.
10. According to the judgment of the investigator, the patients with factors that may affect the results of the study or cause the study to be terminated midway, such as alcoholism, drug abuse, other serious diseases (including mental illness) need to be treated together, severe laboratory abnormalities, accompanied by family or social factors, which will affect the safety of patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  The Objective Response Rate(ORR) is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1.

SECONDARY OUTCOMES:
mORR | 1 year
  The mRECIST Objective Response Rate(mORR) is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by mRECIST.
DOR | 1 year
  The During Of Response(DOR) is defined as the time from the first documentation of CR or PR to the date of first documentation of disease progression as assessed by RECIST 1.1 or death (whichever occurs first).
DCR | 1 year
  The Disease Control Rate(DCR) is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1 .
conversion rate | 1 year
  unresectable converted into resectable
PFS | 1 year
  The progression-free survival time (PFS) defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1 or death, whichever comes earlier.
OS | 1 year
  Overall survival(OS) is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date.
TRAE | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: linhui Peng, Prof, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No